CLINICAL TRIAL: NCT05172661
Title: Effects of Physical-Cognitive Training With Different Task Models on Dual-Task Walking in Parkinson's Disease With Mild Cognitive Impairment
Brief Title: Effects of Physical-Cognitive Training With Different Task Models in Parkinson's Disease With Mild Cognitive Impairment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 202109095RINA
Record Dates: First submitted 2021-11-29; First posted 2021-12-29 (Actual); Last update posted 2023-02-02 (Actual); Status verified 2023-01

CONDITIONS: Mild Cognitive Impairment; Parkinson Disease
Keywords: Dual-task walking training; Parkinson's disease; Mild cognitive impairment; Electroencephalography
MeSH Terms: conditions — Cognitive Dysfunction; Parkinson Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Integrated training model (Experimental): Participants in this group will accept postural and cognitive training at the same time, e.g. naming animals while standing on the foam.
  Each training session will last for 70 minutes, twice a week, and 12 sessions in total.
  Interventions: Behavioral: Integrated physical-cognitive training
- Consecutive training model (Experimental): Participants in this group will accept postural and cognitive training separately and for identical durations (both 30 minutes).
  Each training session will last for 70 minutes, twice a week, and 12 sessions in total.
  Interventions: Behavioral: Consecutive physical-cognitive training

INTERVENTIONS:
Behavioral: Integrated physical-cognitive training — Perform a postural task and a cognitive task at the same time (dual-task model) 70 minutes/session*2 sessions/week*6 weeks
  Arms: Integrated training model
Behavioral: Consecutive physical-cognitive training — Perform a postural task and a cognitive task separately for identical durations 70 minutes/session*2 sessions/week*6 weeks
  Arms: Consecutive training model

SUMMARY:
The present study will characterize exercise model effects (integrated model vs. consecutive model) of physical-cognitive exercise on dual-task walking control in Parkinson's disease with mild cognitive impairment.

ELIGIBILITY:
Inclusion Criteria:

* a diagnosis of idiopathic Parkinson's disease
* have decreased cognitive functions but do not interfere with functional independence
* Montreal Cognitive Assessment (MoCA): 21-25
* able to walk independently without walking devices for at least 10 meters and with the ability to turn 180°

Exclusion Criteria:

* a diagnosis of dementia
* other diseases that may influence cognitive functions or walking performance
* a history of brain surgery
* modification of the medication during the exercise intervention

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2021-11-26 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline dual-task walking performance at 8 weeks | 8 weeks
Fall frequency | 20 weeks
Change from baseline Montreal Cognitive Assessment (MoCA) score at 8 weeks | 8 weeks
  MoCA: 0-30 points, higher scores mean a better outcome

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No